CLINICAL TRIAL: NCT05439577
Title: A Multicentre, Prospective and Registry Study to Explore the Efficacy and Safety of Mucopolysaccharide Polysulfate Cream in the Treatment of Patients With Eczema
Brief Title: A Multicentre Study to Explore the Efficacy and Safety of Mucopolysaccharide Polysulfate Cream in Patients With Eczema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen Kangzhe Pharmaceutical Co., Ltd. (Industry)
Collaborators: Beijing Friendship Hospital (Other); LanZhou University (Other); The First Hospital of Hebei Medical University (Other); Xingtai People's Hospital (Other); Beijing Boai Hospital (Other); Guangxi Ruikang Hospital (Other); The Third Affiliated Hospital of Southern Medical University (Other Government); The Second Affiliated Hospital of Jiaxing University (Other); Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMS-Hirudoid-001
Record Dates: First submitted 2022-06-21; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Eczema
MeSH Terms: conditions — Eczema | interventions — Hirudoid; Glucocorticoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mucopolysaccharide Polysulfate Cream: Prescribed only for patients with Mucopolysaccharide Polysulfate Cream.
  Interventions: Drug: Mucopolysaccharide Polysulfate Cream
- Mucopolysaccharide Polysulfate Cream and glucocorticoids: Patients whose prescriptions contain Mucopolysaccharide Polysulfate Cream and glucocorticoids (Combination therapy, but not always).
  Interventions: Drug: Mucopolysaccharide Polysulfate Cream and glucocorticoids

INTERVENTIONS:
Drug: Mucopolysaccharide Polysulfate Cream — Patients using Hirudoid® alone
  Other Names: Hirudoid®
  Groups: Mucopolysaccharide Polysulfate Cream
Drug: Mucopolysaccharide Polysulfate Cream and glucocorticoids — Patients using Hirudoid® and glucocorticoids (Combination therapy, but not always)
  Other Names: Hirudoid® and glucocorticoids
  Groups: Mucopolysaccharide Polysulfate Cream and glucocorticoids

SUMMARY:
The study was designed to collect information over 1800 patients with a clinical diagnosis of subacute or chronic eczema, these patients' prescriptions contain Hirudoid®. EASI, IGA and more indicators are evaluated. Data were collected for a maximum of 12 weeks according to the clinician's consultation and follow-up (Time points were set at baseline, 1, 2, 3, 4, 8 and 12 weekends). The above data were analysed to explore the optimal treatment modality, dose and treatment period for patients with subacute or chronic eczema.

DETAILED DESCRIPTION:
The study was designed to collect information over 1800 patients with a clinical diagnosis of subacute or chronic eczema, these patients' prescriptions contain Hirudoid® (Hirudoid® alone or in combination with glucocorticoids). Basic demographic information (age, sex, height, weight, lifestyle, occupation), vital signs (blood pressure, heart rate, temperature, etc.), past medical and treatment history, eczema area and severity index (EASI) scores and corresponding symptom scores, Dermatology Life Quality Index (DLQI) score, Investigator's global assessment (IGA) of disease severity score, Visual analogue scale (VAS) with subject's pruritus, photographs of the eczema area and recurrence rate were collected. Data were evaluated for a maximum of 12 weeks according to the clinician's consultation and follow-up (Time points were set at baseline, 1, 2, 3, 4, 8 and 12 weekends). The above data were analysed to explore the optimal treatment modality, dose and treatment period for patients with subacute or chronic eczema.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years of age, male or female;.
2. Patients with a clinical diagnosis of subacute or chronic eczema and whose prescription contains Hirudoid®.
3. Subjects fully understand the content of this study, sign informed consent.

Exclusion Criteria:

1. Hypersensitivity to any of the ingredients of this product.
2. Patients with heparin hypersensitivity, bleeding-prone constitution and known heparin-induced thrombocytopenia.
3. Open wounds and broken skin and mucous membranes
4. Patients with localized combined bacterial, viral and fungal infections.
5. Pregnant or lactating women or those who are unable to use contraception during the study period
6. Those with psychiatric disorders, poor compliance and unable to complete the study.
7. Any other reason that the investigator considers inappropriate for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with subacute or chronic eczema
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
EASI score | It could be any time point in the weekend of 1, 2, 3, 4, 8 and 12
  The greatest change in EASI score occurred during the 12 weeks (follow up point were set at baseline, 1, 2, 3, 4, 8 and 12 weekends) after dosing compared to baseline.

SECONDARY OUTCOMES:
Clinical manifestations. Including Erythema, Thickness (induration, papulation, swelling), Scratching (excoriation), Lichenification (lined skin, furrowing, prurigo nodules). | Baseline, 1, 2, 3, 4, 8 and 12 weekends
  The change in clinical manifestations during treatment compared with at baseline: including Erythema, Thickness (induration, papulation, swelling), Scratching (excoriation), Lichenification (lined skin, furrowing, prurigo nodules).
  Score 0 = no skin lesions, Score 1 = mild, requiring close observation to be seen, Score 2 = moderate, signs visible, Score 3 = severe, signs very visible.
Visual analogue scale (VAS) score | Baseline, 1, 2, 3, 4, 8 and 12 weekends
  The degree of improvement in the subject's self-assessment of visual analogue scale (VAS) compared with that at baseline. The Visual analogue scale (VAS) score was included 11 levels, the minimum value is zero, which means no pruritus; the maximum value is 10, which means extreme pruritus.
The investigator's global assessment (IGA) score | Baseline, 1, 2, 3, 4, 8 and 12 weekends
  The investigator's global assessment (IGA) of disease severity compared to that at baseline. The investigator's global assessment (IGA) score was included 5 levels, the minimum value is zero, which means no eczema-like lesions; the maximum value is 4, which means extremely severe eczema-like lesions.
Recurrence rate. | 8 and 12 weekends
  (Recurrence follow-up on the 8th and 12th weekends is only for patients who have recovered within 4 weeks. Recurrence rate = number of recurrences / number of recovered persons * 100%); Definition of recovery: Subjects with an IGA score of 0 or 1 during the treatment period (within the first 4 weeks).
  Definition of relapse: A recovered patient with an IGA score ≥ 2 at follow-up was judged to be recurred.
Dermatology Life Quality Index (DLQI) score. | Baseline, 1, 2, 3, 4, 8 and 12 weekends
  The Dermatology Life Quality Index (DLQI) score was included 10 questions, each question contains 4 levels, serious (3 score), moderate (2 score), mild (1 score), none or uncorrelated (0 score), respectively. Higher scores indicate greater troubles and annoyances on dermatology life quality from eczema.
Adverse event | 1, 2, 3, 4, 8 and 12 weekends
  Adverse event/serious adverse event was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Lingfeng Li, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China